CLINICAL TRIAL: NCT05869474
Title: Endoscopic Ultrasound-guided Intratumoral Iodine125-Seeds Implantation Combined With Gem/Nab-P Chemotherapy Versus Gem/Nab-P Alone for Metastatic Pancreatic Carcinoma: a Randomized, Controlled, Trial
Brief Title: Implantation of iodine125-Seeds Combined With Chemotherapy in the Treatment of Metastatic Pancreatic Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Department of Gastroenterology, Changhai Hospital, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-219
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: iodine 125; EUS-guided implantation; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Patients will be randomly assigned(1:1) to the two treatment groups by an independent staff who is not involved in the treatment. The endoscopist and patient are not masked because they exactly know whether EUS-guided implantation is performed or not. Survival will be assessed by blinded researchers during follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I125-AG (Experimental): Participants will receive the implantation of radioactive seeds under EUS guide. 48h after implantation, chemotherapy with Gemcitabine 1000mg/m2 plus albumin paclitaxel 125mg/m2 given on days 1 and 8 of each 21-day cycle will be conducted.
  Interventions: Procedure: Iodine125-Seeds implantation; Drug: Gem/nab-P Chemotherapy
- AG (Active Comparator): Participants receive chemotherapy alone. Gemcitabine 1000mg/m2 plus albumin paclitaxel 125mg/m2 given on days 1 and 8 of each 21-day cycle.
  Interventions: Drug: Gem/nab-P Chemotherapy

INTERVENTIONS:
Procedure: Iodine125-Seeds implantation — Endoscopic ultrasound-guided intratumoral iodine125-Seeds implantation
  Arms: I125-AG
Drug: Gem/nab-P Chemotherapy — nab-paclitaxel (125 mg per square meter of body-surface area) followed by gemcitabine (1000 mg per square meter) on days 1, 8 every 3 weeks

SUMMARY:
The goal of this clinical trial is to evaluate the clinical efficacy and safety of endoscopic ultrasonography (EUS)-guided radioactive iodine 125 seeds in combination with AG regimen chemotherapy for the treatment of metastatic pancreatic cancer. The main questions it aims to answer are:

* whether the combination of minimally invasive endoscopy-guided local radiation therapy with chemotherapy may improve overall survival
* the adverse events of the combination therapy Participants will receive the implantation of radioactive seeds under EUS guide. 48h after implantation, chemotherapy with Gem/nab-P given on days 1 and 8 of each 21-day cycle will be conducted.

Researchers will compare the I125+AG group with the group that takes AG chemotherapy alone to see if the overall survival can be improved.

ELIGIBILITY:
Inclusion Criteria:

(Before the trial, subjects must meet all of the requirements listed below in order to be enrolled)

1. 18 to 80 years old;
2. Stage IV pancreatic ductal adenocarcinoma with distant metastases confirmed by clinical, imaging, and pathology, and the primary and metastatic mass can be measured on imaging.
3. No treatment history of chemotherapy, radiotherapy, or surgery
4. Expected survival > 6 months
5. ECGO score of 0-2
6. Eligible for chemotherapy (white blood cell > 3.5×109/L, neutrophil value > 1.5×109/L, hemoglobin > 80g/L, platelets > 100×109/L, albumin > 25g/L, alanine aminotransferase or aspartate aminotransferase ≤ 3 times the upper limit of normal and total bilirubin level ≤ 34.2umol/L, creatinine < 176.8 umol/L, normal ECG)
7. Signed written informed consent;

Exclusion Criteria:

1. Contraindication of EUS-guide procedure or technical infeasibility (e.g.,coagulation disorder, anatomical changes, large vessels along the puncture path)
2. Pregnant or breastfeeding
3. Presence of brain metastases
4. Presence of deep vein thrombosis or pulmonary embolism
5. Presence of HIV, HBV, HCV infection or other uncontrollable active infection
6. Hypersensitivity to chemotherapy drugs
7. History of other malignancies within 5 years
8. Peripheral neuropathy or interstitial lung disease within 5 years
9. Patient is enrolled in any other clinical protocol or investigational trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 48 months
  OS is defined as the time from the date of randomization to the date of death (any cause). Patients who are alive will be censored at the last known time that the patient was alive.

SECONDARY OUTCOMES:
Incidence and severity of Adverse events (AEs) | 48 months
  AEs are graded and reported using The CTCAE version 5.0.
Progression-free survival (PFS) | 48 months
  PFS is defined as the time from the date of randomization to the date of objective disease progression according to RECIST 1.1 criteria or death (due to any cause),whichever occurs first.
Overall Response Rate (ORR) | 48 months
  ORR is defined as the percentage of patients with an investigator-assessed complete (CR) or partial response (PR) according to RECIST v1.1.
CA19-9 response | 48 months
  CA19-9 response is defined as a decrease of CA19-9 concentration by 50% from the prespecified baseline concentration of 74 U/mL or more.
Metabolic response | from baseline to the end of 2nd chemotherapy cycle
  Metabolic response is evaluated by PET/CT according to EORTC criteria.
Visual analog scale (VAS) | 48 months
  Pain is scored according to a VAS score, with a score of 0 indicating no pain and a score of 10 indicating the most intense degree of pain (unbearable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Shen Li, M.D, Principal Investigator — Department of Gastroenterology, Changhai Hospital, Naval Medical University (Second Military Medical University), Shanghai, China.
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No